CLINICAL TRIAL: NCT05234580
Title: A Phase 2 Clinical Study to Evaluate the Safety and Efficacy of PA9159 Nasal Spray for the Treatment of Seasonal Allergic Rhinitis
Brief Title: Safety and Efficacy Study of PA9159 Nasal Spray for the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA9159-201
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PA9159 10 μg (Experimental): Fifty subjects will be randomly assigned to receive 10 μg of PA9159 Nasal Spray for 14 days. Subjects will be administered two vials of drug (spray bottle A and spray bottle B) once daily in the morning, one spray each in the left and right nostril, in the order of first spray A and then spray B. Spray Bottle A: 5 μg/spray; Spray Bottle B: 0 μg/spray.
  Interventions: Drug: PA9159 nasal spray solution, 10 μg once daily for 14 days
- PA9159 20 μg (Experimental): Fifty subjects will be randomly assigned to receive 20 μg of PA9159 Nasal Spray for 14 days. Subjects will be administered two vials of drug (spray bottle A and spray bottle B) once daily in the morning, one spray each in the left and right nostril, in the order of first spray A and then spray B. Spray Bottle A: 0 μg/spray; Spray Bottle B: 10 μg/spray.
  Interventions: Drug: PA9159 nasal spray solution, 20 μg once daily for 14 days
- PA9159 40 μg (Experimental): Fifty subjects will be randomly assigned to receive 40 μg of PA9159 Nasal Spray for 14 days. Subjects will be administered two vials of drug (spray bottle A and spray bottle B) once daily in the morning, one spray each in the left and right nostril, in the order of first spray A and then spray B. Spray Bottle A: 10 μg/spray; Spray Bottle B: 10 μg/spray.
  Interventions: Drug: PA9159 nasal spray solution, 40 μg once daily for 14 days
- Placebo (Placebo Comparator): Fifty subjects will be randomly assigned to receive placebo Nasal Spray without active of PA9159 for 14 days. Subjects will be administered two vials of drug (spray bottle A and spray bottle B) once daily in the morning, one spray each in the left and right nostril, in the order of first spray A and then spray B. Spray Bottle A: 0 μg/spray; Spray Bottle B: 0 μg/spray.
  Interventions: Drug: Placebo nasal spray solution without PA9159, once daily for 14 days

INTERVENTIONS:
Drug: PA9159 nasal spray solution, 10 μg once daily for 14 days — PA9159 of 10 μg is delivered intranasally through a metered-dose mechanical spray pump, once daily in the morning for 14 days.
  Arms: PA9159 10 μg
Drug: PA9159 nasal spray solution, 20 μg once daily for 14 days — PA9159 of 20 μg is delivered intranasally through a metered-dose mechanical spray pump, once daily in the morning for 14 days.
  Arms: PA9159 20 μg
Drug: PA9159 nasal spray solution, 40 μg once daily for 14 days — PA9159 of 40 μg is delivered intranasally through a metered-dose mechanical spray pump, once daily in the morning for 14 days.
  Arms: PA9159 40 μg
Drug: Placebo nasal spray solution without PA9159, once daily for 14 days — Placebo nasal spray solution is delivered intranasally through a metered-dose mechanical spray pump, once daily in the morning for 14 days.
  Arms: Placebo

SUMMARY:
PA9159 is a highly potent novel corticosteroid. The purpose of this study is to evaluate the safety, efficacy and characteristics of population pharmacokinetics of multiple dosing of PA9159 Nasal Spray in patients with seasonal allergic rhinitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel, placebo-controlled clinical trial. Subjects of 200 with seasonal allergic rhinitis are planned to be included in this study. With a ratio of 1: 1: 1: 1 to be randomized allocated to receive PA9159 Nasal Spray of 10 μg, 20 μg, and 40 μg, or placebo, with 50 subjects in each group. The duration of this study is approximately 12 months, including screening, baseline, treatment observation, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years, male or female;
* Clinical diagnosis is based on the Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2018 Edition) issued by the Rhinology Group of the Otorhinolaryngology Head and Neck Surgery Branch of the Chinese Medical Association, with a clear history of Seasonal Allergic Rhinitis (SAR) ≥ 1 year (written or verbal confirmation), and positive test for one or more allergens before randomization. Recognize the results of any one of the skin prick test (SPT), intradermal test, and serum specific IgE test; Clinical manifestations may include:

  1. Symptoms: 2 or more symptoms such as sneezing, runny nose, itchy nose and nasal congestion, lasting or accumulating for more than 1 h each day, may be accompanied by ocular symptoms such as itching, lacrimation, and red eyes;
  2. Signs: pallor and edema of the nasal mucosa and watery nasal secretions;
  3. Allergic symptoms are characterized by seasonal onset in spring and/or fall, and at the time of this enrollment, it is during the onset of symptoms.
* Reflective Total Nasal Symptom Score (rTNSS) ≥ 6 points, nasal congestion ≥ 2 points, and one of the three symptoms of sneezing, runny nose and itchy nose ≥ 2 points, all these three conditions are met simultaneously at the time of screening, baseline and the first dosing during treatment; The mean rTNSS at baseline was the mean of a total of 8 scores on evening of D-4, morning and evening of D-3, D-2 and D-1, and the morning of D1;
* Capable of demonstrating the correct use of nasal spray techniques after training at screening;
* Capable of performing respiratory exercise as required at the time of intranasal administration after training at screening;
* Is willing to sign the informed consent form (ICF), comply with the study procedures, including the correct use of the nasal spray device, and understand and accurately record the patient diary card; Ability to understand and receive treatment, laboratory tests, and other study procedures as planned.

Exclusion Criteria:

* Previous intolerance to intranasal administration;
* Patients with asthma requiring long-term treatment (patients with occasional acute asthma, or mild, exercise-induced asthma requiring no medication or only beta-agonist treatment during the study may be included);
* Active or inactive tuberculosis infection, untreated local or systemic fungal, bacterial, viral, or parasitic infection;
* Presence of glaucoma, cataract, ocular herpes simplex, infectious conjunctivitis, or other ocular infections (except allergic conjunctivitis);
* Any nasal mucosal erosion, septal ulceration, or nasal septal perforation at screening or prior to the first dose on D1;Presence of other nasal disorders that may affect intranasal drug deposition as judged by the investigator, such as acute or chronic sinusitis, drug-induced rhinitis, nasal polyps, or nasal septal deviation;
* History with sinus surgery within 3 months or nasal trauma that have not completely healed;
* Respiratory tract infections treated with antibiotics within 4 weeks prior to screening;
* Patients with severe lung diseases, such as COPD (chronic obstructive pulmonary disease), etc.;
* Patients with unstable heart disease with drug-control;
* Patients who have received desensitization therapy within 6 months prior to screening;
* Severe liver and kidney disease, or abnormal liver and kidney function tests (ALT, AST ≥ 2 times the upper limit of normal, or Cr > 1.2 times the upper limit of normal);
* Use of short-lasting prescriptions and OTC antihistamines within 3 days prior to screening; Use of nasal glucocorticoids within four weeks; Inhalation, oral, intramuscular/intravascular injection, topical hormones (except hydrocortisone cream containing ≤ 1%) within 8 weeks prior to screening; Use of nasal or ophthalmic cromoglycic acid within 14 days prior to screening; Use of long-lasting antihistamines such as loratadine, desloratadine, fexofenadine, or cetirizine within 10 days prior to screening; Oral or nasal decongestants, nasal anticholinergics, or oral antileukotrienes within 72 h prior to screening; Use of Omalizumab subcutaneously within 5 months prior to screening; Use of anti-allergic Chinese herbal medicines within 14 days prior to screening.
* Planned use of the following medications or/and treatments during the study: a. Strong CYP3A4 inhibitors, such as ketoconazole, clarithromycin, etc.; b. Chronic or intermittent use of inhaled, oral, intramuscular, intravenous, and/or potent topical corticosteroids; c. Antihistamines (except salvage medications required during the trial); d. Leukotriene modulators; e. Mast cell membrane stabilizers (including cromoglycate sodium, nidolate sodium, tetrazolone, nedocromil sodium, pemirolast potassium, and tranilast, etc.); f. Decongestants; g. Anticholinergics; h. Immunotherapeutic agents; i. Anti-allergic Chinese herbal medicine;
* Planned to travel outside the local area for 2 consecutive days (48 h) or a total of more than 3 days during the trial;
* Alcohol addicts in the previous 1 year (alcoholism defined as: greater than 14 units of alcohol per week;1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits or 150 mL of wine containing 40% alcohol), drug abusers, drug addicts, or smoking addicts (average of more than 10 cigarettes per day);
* Allergic to the investigational drug and its excipients;
* Pregnant or lactating women, and male subjects (or their partners) or female subjects who have a pregnancy plan throughout the trial and for 3 months after the end of the study;
* Participated in other drug clinical trials within 3 months prior to screening, and used the study drug;
* Based on the judgment of the investigator, the subject may have an impact on compliance with any aspect of the protocol (including visit plan and completion of diary cards or questionnaires) due to physical, educational level, or geographic location;
* Based on the opinion of the investigator, there are any circumstances that may affect the subject's informed consent or compliance with the protocol, or that the subject's participation in the trial may affect the results of the study or their own safety.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Evaluation the change from baseline in daily subject-reported AM and PM Reflective Total Nasal Symptom Score (rTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Nasal Symptom Score (rTNSS) measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.

SECONDARY OUTCOMES:
Evaluation the proportion and frequency of patients using the antihistamine drug of loratadine tablets during the treatment period; | From pre-dose until 14 days post-dose
  If the subject is intolerant of symptoms, loratadine tablets may be taken with the consent of the investigator, 10 mg once a day, without overdose; If symptoms improve, they will no longer be used; It can be used once or continuously for ≤ 3 days, preferably avoiding intermittent use. Continue study drug while taking salvage medication.
Evaluation the change from baseline in daily subject-reported AM and PM Instantaneous Total Nasal Symptoms Scores (iTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. mild
  2. moderate
  3. severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Instantaneous Total Nasal Symptoms Scores (iTNSS) measures these symptoms over the previous 10 minute time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the Area Under the Curve (AUC) of Reflective Total Nasal Symptom Score (rTNSS) over time in subjects. | From pre-dose until 14 days post-dose
  The parameter of AUC was produced based on the Reflective Total Nasal Symptom Score (rTNSS) obtained daily over the 14-day treatment period.
Evaluation the change from baseline in subject-reported Instantaneous Total Nasal Symptoms Scores (iTNSS) at 4 h ± 0.5 h, 8 h ± 0.5 h, and 12 h ± 1 h after the first dose in the treatment period. | Day 1 of the first dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. mild
  2. moderate
  3. severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Instantaneous Total Nasal Symptoms Scores (iTNSS) measures these symptoms over the previous 10 minute time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline in daily subject-reported AM Reflective Total Nasal Symptom Score (rTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Nasal Symptom Score (rTNSS) measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline in daily subject-reported PM Reflective Total Nasal Symptom Score (rTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Nasal Symptom Score (rTNSS) measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the percentage change from baseline in subject-reported AM and PM Reflective Total Nasal Symptom Score (rTNSS) averaged on a subject-day basis. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Nasal Symptom Score (rTNSS) measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the percentage change from baseline in daily subject-reported AM Instantaneous Total Nasal Symptoms Scores (iTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Instantaneous Total Nasal Symptoms Scores (iTNSS) measures these symptoms over the previous 10 minute time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the percentage change from baseline in daily subject-reported PM Instantaneous Total Nasal Symptoms Scores (iTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Instantaneous Total Nasal Symptoms Scores (iTNSS) measures these symptoms over the previous 10 minute time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the percentage change from baseline in daily subject-reported AM Reflective Total Nasal Symptom Score (rTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Nasal Symptom Score (rTNSS) measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the percentage change from baseline in daily subject-reported PM Reflective Total Nasal Symptom Score (rTNSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Nasal Symptom Score (TNSS) is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, Total Nasal Symptom Score (TNSS) values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Nasal Symptom Score (rTNSS) measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline in overall score of the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) in participants over the 14-day treatment period. | From pre-dose until 14 days post-dose
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28).
  Therefore, Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) values range from 0-168 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline in overall score of the Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) in participants over the 14-day treatment period. | From pre-dose until 14 days post-dose
  The Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) has 16 items in 4 domains (problems with sleep, symptoms during sleep time, symptoms on waking in the morning and practical problems). Each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Patients recall their experiences during the previous week and respond to each question.
  Therefore, Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) values range from 0-96 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline in daily subject-reported AM and PM Reflective Total Ocular Symptom Score (rTOSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Ocular Symptom Score (TOSS) is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. mild
  2. moderate
  3. severe Therefore, Total Ocular Symptom Score (TOSS) ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Reflective Total Ocular Symptom Score (rTOSS) symptom scores assess symptoms over the previous 12-hour time interval. Difference was calculated as 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline in daily subject-reported AM and PM Instantaneous Total Ocular Symptoms Scores (iTOSS) averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  Total Ocular Symptom Score (TOSS) is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. mild
  2. moderate
  3. severe Therefore, Total Ocular Symptom Score (TOSS) ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  The parameter of Instantaneous Total Ocular Symptoms Scores (iTOSS) symptom scores assess symptoms over the previous 10 minute time interval. Difference was calculated as 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Evaluation the change from baseline of each individual rhinitis symptom score averaged over the 14-day treatment period. | From pre-dose until 14 days post-dose
  The individual rhinitis symptoms are runny nose, sneezing, itchy nose, and nasal congestions. Difference was calculated as the 14-day treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, phD, Principal Investigator — Beijing Tongren Hospital
Locations (17):
- China (17):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing TongRen Hospital, Beijing, Beijing Municipality
  - Dongfang Hospital Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Yanbian University Hospital(Yanbian Hospital), Yanji, Jilin
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No